CLINICAL TRIAL: NCT06433284
Title: Comparative Study of Decellularized Human Amniotic Membrane Hydrogel and Inverted Internal Limiting Membrane Flap in Idiopathic Large Macular Holes (MACROHOLE): a Randomized-control Trial
Brief Title: Comparative Study of Decellularized Human Amniotic Membrane Hydrogel and Inverted Internal Limiting Membrane Flap in Idiopathic Large Macular Holes
Acronym: MACROHOLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Walailak University (Other)
Responsible Party: Principal Investigator, Jakkrit Juhong, Head of Vitreoretinal unit, Ophthalmology department, Walailak University, Walailak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WU999
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Macular Holes
Keywords: macular holes; decellularized amniotic membrane; human amniotic membrane hydrogel
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inverted flap (Active Comparator): Patients who will undergo 25-gauge pars plana vitrectomy with inverted flap technique and SF6 tamponade.
  Interventions: Procedure: 25-gauge pars plana vitrectomy with inverted flap technique and SF6 tamponade
- Amniotic membrane hydrogel (Experimental): Patients who will undergo 25-gauge pars plana vitrectomy with complete internal limiting membrane peeling, amniotic membrane hydrogel filling and SF6 tamponade.
  Interventions: Procedure: 25-gauge pars plana vitrectomy with complete internal limiting membrane peeling with amniotic membrane hydrogel filling and SF6 tamponade

INTERVENTIONS:
Procedure: 25-gauge pars plana vitrectomy with inverted flap technique and SF6 tamponade — Standard 3 port 25-gauge pars plana vitrectomy with inverted flap technique after brilliant blue dye staining and SF6 tamponade. "Flower petal" type of inverted flap will be performed - multiple small ILM flaps will be created around the macular hole and placed over the macular hole
  Arms: Inverted flap
Procedure: 25-gauge pars plana vitrectomy with complete internal limiting membrane peeling with amniotic membrane hydrogel filling and SF6 tamponade — Standard 3 port 25-gauge pars plana vitrectomy with complete internal limiting membrane peeling around the macular hole after brilliant blue dye staining then filling the hole with amniotic membrane hydrogel and sulfur hexafluoride (SF6) tamponade
  Arms: Amniotic membrane hydrogel

SUMMARY:
The human amniotic membrane (hAM) patch, introduced by Rizzo et al. in 2018, showed a 100% anatomical success rate for large or failed macular holes over a 6-month follow-up. Despite its regenerative properties like promoting angiogenesis and having low immunogenicity, its clinical use is limited by challenges such as trimming to fit small holes and complications during insertion. To overcome these issues, decellularized amniotic membrane (dAM) has been processed into a hydrogel form, enhancing its applicability and allowing it to be used as an injectable hydrogel for minimally invasive therapies. While dAM hydrogels have been used in various medical fields, their application in intraocular surgery is new. This study proposes using dAM hydrogel for large macular hole closure, comparing its effectiveness to the inverted ILM flap technique in a randomized controlled trial.

DETAILED DESCRIPTION:
A macular hole (MH) is a neuroepithelial defect in the macular area of the retina. The estimation of macular hole incidence about 33 of every 10,000 person in individuals older than 55 years old1. The female-to-male ratio is 2 to 3:1. Idiopathic macular hole (IMH) is MHs occurring independently of primary ocular diseases such as trauma and vitreoretinopathy2 and represents the predominant subtype of MH, constituting approximately 83%1. There is a 5% to 15% risk of developing macular hole in the other eye if a macular hole develops in one eye.1 In 1988, Gass proposed a classification system for idiopathic macular holes, as well as a new hypothesis for its pathogenesis, which emphasizes the role of the vitreo-macular tangential traction in the formation of macular holes3. Macular hole closure can occurred spontaneously in approximately 5-10% cases in early stages. Pars plana vitrectomy with internal limiting membrane (ILM) peeling and gas tamponade has been the standard of care of small size macular hole treatment with success rate more than 90%4. However, in large macular hole more than 400 um, the success rate is lower. Previous study showed closure rate of large macular hole > 400 μm is 56% with poor visual outcome.4,5 Several new techniques have been described to improve anatomical and functional outcomes in cases of large macular holes by inserting alternative tissues into the macular hole, such as the ILM flap, human amniotic membrane patch6, or retinal tissue implantation, to promote anatomical closure and improve visual acuity. The utilization of ILM flap coverage has emerged as an effective surgical approach for treating large, full-thickness idiopathic MH and myopic MH. This technique was initially introduced in 1999, showing promising results in enhancing macular hole closure rates through ILM peeling. Several subsequent studies 7-9 have further substantiated the efficacy of ILM flap coverage, making it the standard surgical treatment for large macular hole cases. However, this technique is often hindered by limitations related to the technical complexity of surgery and the risk of retinal trauma.

The human amniotic membrane (hAM) patch, proposed by Rizzo et al. in 20186, serves as another alternative technique for large or failed macular hole cases. The anatomical success rate was 100% during the 6 months follow-up. The exceptional biological properties of hAM, including its promote angiogenesis10, low immunogenicity11, and anti-inflammatory11,12, anti-fibrotic13, and antibacterial characteristics14, make it highly suitable for regenerative medicine and intraocular implantation. However, the clinical application of thin hAM sheets is limited by several challenges, such as the difficulty of trimming it to fit very small hole sizes (< 0.2 cm), tissue loss after insertion into the PPV port, and complications during the insertion of the hAM patch into the hole. To address these limitations, processing decellularized amniotic membrane (dAM) tissue into a hydrogel form has enhanced its processability and applicability15. This transformation allows it to be used as an injectable hydrogel for minimally invasive therapies and facilitates its manipulation into the macular hole.

dAM hydrogels have been applied in various fields, including skin repair, cardiac treatment, cartilage regeneration, endometrial regeneration, vascular grafts, dental pulp regeneration, and as cell culture/carrier platforms. However, their use in intraocular surgery has not yet been established. Additionally, the benefits of dAM hydrogel over hAM tissue include lower immunogenicity due to the decellularization processs since the resident cells may cause intense host immunologic reactions after transplantation and transplant rejection and the homogeneous distribution of biochemical substances within the hydrogel structure.15 In this study, we will be the first to propose a new technique and invention for closing large macular holes using human amniotic membrane hydrogel filling in the hole after standard ILM peeling. We conducted a randomized controlled trial to compare the anatomical and visual outcomes of the inverted ILM flap technique (IFT) with the dHM hydrogel technique in idiopathic large macular holes with a minimum diameter (MD) greater than 400 μm.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* idiopathic full thickness macular hole > 400 micron of diameter
* phakic or pseudophakic
* absence of systemic adverse conditions

Exclusion Criteria:

* idiopathic full thickness macular hole > 1,500 micron of diameter
* traumatic macular holes
* myopic macular holes,
* concomitant retinal and other ocular disease
* previous ocular surgery except cataract surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | 6 months
  Difference of best corrected visual acuity (BCVA) after primary vitrectomy for idiopathic full thickness macular holes with inverted flap technique versus internal limiting membrane (ILM) peeling technique
Closure rate | 6 months
  Closure rate after primary vitrectomy for idiopathic full thickness macular holes with decellularized amniotic membrane hydrogel versus inverted flap technique

CONTACTS AND LOCATIONS:
Overall Officials: Jakkrit Juhong, MD., Principal Investigator — School of Medicine, Walailak university